CLINICAL TRIAL: NCT05140642
Title: Blinded Randomized Controlled Trial of Artificial Intelligence Guided Assessment of Cardiac Function
Brief Title: Safety and Efficacy Study of AI LVEF
Acronym: EchoNet-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, David Ouyang, Staff Physician, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: STUDY00001707
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure, Systolic; Heart Failure, Diastolic
Keywords: Echocardiogram; Artificial Intelligence
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure, Diastolic

STUDY DESIGN:
Intervention Model Description: Studies will be randomized 1:1 to either sonographer preliminary report finding or AI preliminary report finding with final adjudication by the cardiologist. With AI preliminary report, the preliminary interpretations will be generated by AI (artificial intelligence) technology [a semantic segmentation model] and the PACS system's native EF calculation workflow will be used to calculate LVEF. The study team will assess how much cardiologists edit and change this preliminary interpretation is from the final interpretation.
Who Masked: Participant
Masking Description: Measurements shown in Picture Archiving and Communication System (PACS) without direct communication between sonographer and cardiologist. Annotations are shown without identifiers on how the annotations were done. Cardiologists are blinded to source of preliminary interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonographer Annotation (Active Comparator): Currently, sonographer technicians provide preliminary interpretations prior to validation and overreading by cardiologists. This staggered, stepwise evaluation allows for the introduction of AI decision support with minimal impact on patient care. Physicians are already used to adjusting the preliminary report given the variable training of sonographers and on the lookout for changes, variation, or adjustments that need to be made.
  Interventions: Other: Sonographer Measurement of LVEF
- Artificial Intelligence Annotation (Experimental): In preliminary work, a novel AI algorithm developed to assess LVEF was shown to be more precise than human interpretation in 10,030 echocardiograms done at Stanford University (Ouyang et al. Nature, 2020). With randomization, a proportion of the preliminary interpretations will be done by AI technology and the study team will assess how different this preliminary interpretation is from the final interpretation.
  Interventions: Other: Automated annotation of the left ventricle through deep learning

INTERVENTIONS:
Other: Automated annotation of the left ventricle through deep learning — A semantic segmentation deep learning model will identify the left ventricle and label the left ventricle. The AI model will produce an assessment of LVEF using video based features.
  Arms: Artificial Intelligence Annotation
Other: Sonographer Measurement of LVEF — Standard practice sonographer measurement of left ventricle and assessment of LVEF
  Arms: Sonographer Annotation

SUMMARY:
To determine whether an integrated AI decision support can save time and improve accuracy of assessment of echocardiograms, the investigators are conducting a blinded, randomized controlled study of AI guided measurements of left ventricular ejection fraction compared to sonographer measurements in preliminary readings of echocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* The study imaging studies will include patients who underwent imaging (limited or comprehensive transthoracic echocardiogram studies) and a LVEF was adjudicated in the echocardiography/non-invasive cardiac imaging laboratory.
* The study participants are cardiologists reading in the echocardiography/non-invasive cardiac imaging laboratory.

Exclusion Criteria:

* The study imaging studies will exclude transesophageal echocardiogram imaging.
* The study will exclude cardiologists who decline to participate

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3495 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Frequency of >5% change in LVEF between preliminary and final report | 10 Minutes
  Proportion of studies the LVEF is changed more than 5% in final report
Average change in LVEF between preliminary and final report | 10 Minutes
  Mean change in LVEF between preliminary and final report

SECONDARY OUTCOMES:
Frequency cardiologist adjusts preliminary annotation | 10 Minutes
  Proportion of studies the annotation is changed
Average change in LVEF between prior clinical report and final report | 10 Minutes
  Mean change in LVEF between prior clinical report and final report

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ouyang D, He B, Ghorbani A, Yuan N, Ebinger J, Langlotz CP, Heidenreich PA, Harrington RA, Liang DH, Ashley EA, Zou JY. Video-based AI for beat-to-beat assessment of cardiac function. Nature. 2020 Apr;580(7802):252-256. doi: 10.1038/s41586-020-2145-8. Epub 2020 Mar 25. PMID 32269341
- [Derived] He B, Kwan AC, Cho JH, Yuan N, Pollick C, Shiota T, Ebinger J, Bello NA, Wei J, Josan K, Duffy G, Jujjavarapu M, Siegel R, Cheng S, Zou JY, Ouyang D. Blinded, randomized trial of sonographer versus AI cardiac function assessment. Nature. 2023 Apr;616(7957):520-524. doi: 10.1038/s41586-023-05947-3. Epub 2023 Apr 5. PMID 37020027